CLINICAL TRIAL: NCT04372576
Title: Epidemiology and Outcome of Ventilator-associated Pneumonia Among Critically Ill COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Zsolt Iványi, Associate Professor, Semmelweis University
Other Study IDs: 57/2020.
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Ventilator Associated Pneumonia; Corona Virus Infection
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of ventilator-associated pneumonia criteria — Diagnosis of ventilator-associated pneumonia is based upon the routine daily clinical and laboratory parameters.

SUMMARY:
The aim of this study is to determine the risk factors for development of ventilator-associated pneumonia (VAP) and to identify the prognostic factors of VAP among Coronavirus Disease 2019 (CoViD-19) patients. We hypothesized that CoViD-19 serves as a high risk factor for the development of VAP and it affects clinical outcome measures negatively.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (CoViD-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) became a pandemic affecting thousands of individuals worldwide. A considerable proportion of CoViD-19 patients require admission to the intensive care unit (ICU), although limited data are available on their clinical characteristics and course. The results of retrospective studies indicate older age, presence of comorbidies and secondary infections as predictors of mortality among this population. Further evaluation regarding ICU clinical course and predictors of mortality is needed.

The aim of this study is to determine the risk factors for development of VAP and to identify the prognostic factors of VAP among CoViD-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill individuals diagnosed with PCR confirmed CoViD-19 disease
* Started mechanical ventilation for > 48 hours
* Informed consent signed by the patient or authorised representative

Exclusion Criteria:

* Participation in an interventional trial aiming nosocomial infections
* refused informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill individuals diagnosed with PCR confirmed CoViD-19 disease requiring mechanical ventilation for > 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | at study completion, anticipated 5 months

SECONDARY OUTCOMES:
Days of mechanical ventilation | average time frame expected 2-3 weeks
ICU length-of-stay | average time frame expected 3-4 weeks
Antibiotic utilization | average time frame expected 3-4 weeks (at discharge from ICU)
Ventilator-associated pneumonia rate | at study completion, anticipated 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No